CLINICAL TRIAL: NCT01402323
Title: A Prospective Split-mouth Designed Study on the Incidence of Gingival Clefts During Orthodontic Space Closure Into Recent or Healed Extraction Sockets.
Brief Title: Gingival Clefts and Orthodontic Movement
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Allocation: Randomized | Masking: Single | Purpose: Treatment
Other Study IDs: EK Nr 105/2011
Record Dates: First submitted 2011-07-25; First posted 2011-07-26 (Estimated); Last update posted 2014-05-20 (Estimated); Status verified 2011-07

CONDITIONS: Gingival Clefts; Extraction Socket; Orthodontic Movement

STUDY DESIGN:
Who Masked: Investigator

ARMS (1):
- early or late tooth extraction (Other)
  Interventions: Other: time point of tooth extraction

INTERVENTIONS:
Other: time point of tooth extraction

SUMMARY:
Clefts or invaginations of the gingival tissue are a frequent finding during orthodontic space closure after extraction of a tooth. They occur in about 35% of the cases. Increased risk of developing a gingival cleft is given in the mandibular arch. A gingival invagination impairs aesthetics, orthodontic treatment and periodontal health. The aim of this prospective split-mouth designed observer blinded study is to evaluate possible differences between tooth movement in recent or in healed extraction sockets on incidence of gingival clefts. We hypothesize, that similar to the results originated from an animal study immediate movement in extraction sockets reduces incidence of gingival clefts during orthodontic space closure.

ELIGIBILITY:
Inclusion Criteria:

* extraction of both molars or premolars in the upper or lower jaw and orthodontic space closure

Exclusion Criteria:

* periodontal status not allowing orthodontic treatment

Min Age: 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2011-07; Primary Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
incidence of gingival clefts | up to 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Bernhard Gottlieb School of Dentistry, Medical University of Vienna, Vienna, Austria